CLINICAL TRIAL: NCT04614181
Title: The Feasibility and Benefits of Pre-operative Whey-protein Infused Carbohydrate Loading in Elderly With Hip Fractures Undergoing Surgery: a Pilot Study
Brief Title: Protein and Carbohydrate Loading in Elderly With Hip Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020629-8833 56379
Record Dates: First submitted 2020-10-20; First posted 2020-11-03 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Hip Fractures
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Carbohydrate and protein loading (Experimental): Nestle Resource drink
  Interventions: Dietary Supplement: Nestle Resource drink
- Usual care (Active Comparator): Usual fracture care as determined by clinical team
  Interventions: Other: Usual care

INTERVENTIONS:
Dietary Supplement: Nestle Resource drink — Beverage (Nestle RESOURCE). Each serving is 237ml containing 53.6g of carbohydrate and 9g of protein. Intervention group will consume two servings of the carbohydrate beverage (53.6g each, total of approximately 100g) on the day before surgery and one serving up to 6 hours prior to scheduled surgery time.
  Arms: Carbohydrate and protein loading
Other: Usual care — Usual fracture care as determined by clinical team
  Arms: Usual care

SUMMARY:
Pre-operative carbohydrate and protein loading among older people with hip fractures could potentially influence patient outcomes. This mode of intervention has seen good outcomes in a general surgical setting as part of its enhanced recovery pathway. However, its effectiveness and ease of implementation in a hip fracture setting is uncertain. This study aims to study the feasibility of protein and carbohydrate loading as part of hip fracture management compared to usual care.

DETAILED DESCRIPTION:
INTRODUCTION AND BACKGROUND

Pre-operative carbohydrate loading is one of the many components of enhanced recovery after surgery (ERAS) protocol. It has been identified as one of the independent predictors among ERAS components to improve peri-operative well-being and reduce post-operative complications. While well-being is a subjective outcome, several surrogate outcomes have been used to quantify some of the aspects. These surrogate outcomes of well-being include post-operative nausea and vomiting, pain, and preservation of muscle strength.

Although the exact mechanism of how pre-operative carbohydrate loading improves these outcomes is unclear, there appears to be an anabolic effect by increasing insulin sensitivity, improving glucose control and reducing catabolism. Patients in anabolic state undergo less post-operative nitrogen and protein loss, which translates to preservation of muscle strength. Carbohydrate loading keeps the body in a fed state during the fasting period before surgery. This abolishes the starvation effects which causes reduced insulin sensitivity commonly seen with conventional fasting practice. This is an independent predictor which prolongs length of hospital stay, preservation of muscle mass and handgrip strength post-operatively.

While most studies have demonstrated benefits of carbohydrate loading in patients undergoing abdominal surgeries, the number of studies conducted in the orthopedic hip fracture population are limited. In addition, there may also be barriers to introducing a new protocol with carbohydrate loading to replace the existing conventional fasting practice. Studies showed diverse feasibility in terms of implementation, which seemed to be multifactorial. More studies are therefore required to identify the factors promoting or impeding such a practice in respective centres. Given that a significant number of the hip fracture population are malnourished elderly who may benefit from this intervention, the gap in literature in this population deserves a thorough attention.

The University Malaya Medical Centre is a tertiary hospital with an average of 200 hip fracture cases annually. To date, these cases are subjected to conventional fasting starting from midnight. They are usually fasted up to extended hours, putting them in a starved state before surgery. It is therefore the great interest of the current multidisciplinary teams involved in the clinical care of hip fracture patients to introduce carbohydrate loading as part of the fasting practice. This study aims to introduce the concept and assess the feasibility of such a practice. The results from this pilot study may be used to revolutionize the fasting practice in our hospital.

OBJECTIVE

Primary objective

1. To study the feasibility of implementing pre-operative carbohydrate loading in patients undergoing hip surgery
2. To study the safety of pre-operative carbohydrate loading in patients undergoing hip surgery

Secondary objective

1. To evaluate the effect of pre-operative carbohydrate loading among patients undergoing hip fracture surgery

METHODS

This is a pilot study to collect data on feasibility of implementing carbohydrate loading before orthopaedic hip fracture surgery. It is also an open labelled, randomized controlled study to identify correlation between pre-operative carbohydrate loading and surrogate outcomes of well-being. A computer generated randomization method will be used to allocate participants to each arm (intervention vs control) on a 1:1 ratio basis. The randomization allocation will be revealed after consent and baseline assessment.

The amount of carbohydrate load required to induce an effect must be enough to shift the body from a fasted to a fed state. A 50g oral carbohydrate ingestion has been shown to stimulate insulin release resembling post-prandial state. Therefore, the ERAS society recommendation is based on the following dose: a loading dose of 100g carbohydrate the day before surgery (as glycogen store) followed by a 50g dose 2 hours before surgery (to keep patients in a fed state).

In our study, the intervention group will receive the carbohydrate beverage (Nestle RESOURCE). Each serving is 237ml containing 53.6g of carbohydrate and 9g of protein. Intervention group will consume two servings of the carbohydrate beverage (53.6g each, total of approximately 100g) on the day before surgery and one serving 6 hours prior to scheduled surgery time. The control group will receive usual hip fracture care as determined by the clinical team.

SAMPLE SIZE

For this pilot study, a sample size of 40 is targeted. 20 will be randomized to the intervention group receiving the supplement drink, while 20 will be randomized to the control group who will not be receiving any supplements. No formal sample size calculation was used. One of the objectives of this feasibility study is to provide estimates of recruitment and retention rates for a larger study. The number of participants for this study will be determined by resources and the recruitment period.

ANALYSIS

Baseline demographic data will be presented as mean ± SEM. Feasibility outcomes will be reported as numbers and percentages. Descriptive statistics (mean, standard deviation, and median for continuous variables; frequencies and percentages for categorical variables) will be calculated separately by group. For the group comparison, appropriate tests based on their distribution will be performed.

ELIGIBILITY:
Inclusion Criteria:

* All patients planned for semi-emergency hip surgery (total arthroplasty, hemiarthroplasty, internal fixation)
* Aged 65 years and above
* ASA 1-3 (ASA Physical Status Classification System)

Exclusion Criteria:

* Patients undergoing hip surgery of emergency nature (inadequate time for recruitment and pre-operative intervention)
* Peri-prosthetic hip fracture and fracture due to underlying malignancy
* Revision hip surgery
* Participation in another nutritional program
* Diabetes mellitus
* Intolerance to carbohydrate drinks
* Gastric reflux, risk of aspiration, dysphagia
* Severe cognitive impairment and delirium

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 34 (Actual)
Dates: Start 2020-11-04 (Actual); Primary Completion 2021-06-29 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
The number of participants recruitment | 6 months
  How many participants willing to be recruited, screening to recruitment rate
The number of participants that adhered to nutritional loading | 6 months
  How many participants adhered to the the total treatment drinks
The attrition rate of participants recruited into the study | 6 months
  How many participants dropped out or had missing data
Safety profile: How many participants had an adverse reaction | 6 months
  How many participants had an adverse reaction

SECONDARY OUTCOMES:
Prevalence of post-operative nausea and/or vomiting | 6 months
  Number of participants with post-operative nausea and/or vomiting
Severity of post-operative pain | 6 months
  Resting and dynamic pain assessed at 48-72 hours
Length of stay | 6 months
  Inpatient length of acute hospital stay
Change in muscle strength | 6 months
  Difference of hand grip strength and anthropometric measurements pre- and post-operatively
Prevalence of post-operative complications | 6 months
  Number of participants that developed complications after surgery (infection, cardiovascular, kidney injury, stroke, thromboembolism, pressure ulcer)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, University of Malaya, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yap KS, Loh PS, Foong YX, Mok CZ, Ong T, Khor HM. A feasibility study on preoperative carbohydrate loading in older patients undergoing hip fracture surgery. BMC Geriatr. 2024 May 6;24(1):401. doi: 10.1186/s12877-024-04958-7. PMID 38711010